CLINICAL TRIAL: NCT02047695
Title: Women With Migraine With Aura Neuroimaging (WOMAN) Study: A Population-based Study of Danish Twins
Brief Title: Women With Migraine With Aura Neuroimaging Study
Acronym: WOMAN
Status: Completed | Type: Observational
Sponsor: Odense University Hospital (Other)
Collaborators: Glostrup University Hospital, Copenhagen (Other); Copenhagen University Hospital, Hvidovre (Other); University of Southern Denmark (Other)
Responsible Party: Principal Investigator, David Gaist, professor, consultant, Odense University Hospital
Other Study IDs: S-20100126
Record Dates: First submitted 2014-01-26; First posted 2014-01-28 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-04

CONDITIONS: Migraine With Aura
Keywords: migraine with aura; migraine; case-control study; magnetic resonance imaging; brain diseases
MeSH Terms: conditions — Migraine with Aura; Migraine Disorders; Brain Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Migraine with aura: Participants with migraine with aura (cases), their co-twins, and unrelated migraine-free twins (controls)

SUMMARY:
The purpose of this study is to investigate whether a particular form of migraine, migraine with aura, is associated with structural changes in the brain

ELIGIBILITY:
Inclusion Criteria:

* female
* case (migraine with aura), co-twin to case, or control (migraine-free)
* residency in Denmark
* no severe neurological (vascular, neurodegenerative or neuroinflammatory) disorders, or other somatic or psychiatric disorders

Exclusion Criteria:

* male
* residency outside Denmark
* registered in Civil Registry as not to be contacted by researchers
* severe neurological (vascular, neurodegenerative or neuroinflammatory) disorders, or other somatic or psychiatric disorders
* mobile metal parts or other contraindication for MRI
* weight of 130+ kilograms
* pregnancy
* subjects that wished not to be informed about abnormal findings on MRI
* chronic tension-type headache, medication overuse headache, or cluster headache (diagnosed through physician interview)
* frequent tension-type headache (control group only, self-reported or diagnosed through physician interview)

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Selected from a population-based twin registry
Sampling Method: Non-Probability Sample
Enrollment: 345 (Actual)
Dates: Start 2011-02; Primary Completion 2015-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Evidence of white matter hyperintensities or subclinical ischaemic stroke confirmed by MRI | At time of MRI

SECONDARY OUTCOMES:
Evidence of other structural and functional changes in brain | At time of MRI

CONTACTS AND LOCATIONS:
Overall Officials: David Gaist, MD, PhD, Principal Investigator — Department of Neurology, Odense University Hospital